CLINICAL TRIAL: NCT06657794
Title: Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Juxtarenal Aortic Aneurysms
Brief Title: Physician Modified Endovascular Grafts for the Treatment of Juxtarenal Aortic Aneurysms
Acronym: PMEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Sean Lyden, MD, Sponsor-Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-009
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Juxtarenal Aortic Aneurysm; Aortic Rupture
MeSH Terms: conditions — Aortic Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention (Experimental): Implantation of Physician-Modified Terumo Aortic TREO abdominal stent graft system
  Interventions: Device: Implantation of Physician-Modified Terumo Aortic TREO abdominal stent graft system

INTERVENTIONS:
Device: Implantation of Physician-Modified Terumo Aortic TREO abdominal stent graft system — A Physician Modified Endograft is a commercially available, off-the-shelf endograft that has been altered at the time of the procedure by creating fenestrations in the seal zone of the graft to preserve blood flow into vital branch vessels. These fenestrations are marked with medical grade gold markers to facilitate fluoroscopic visualization during the procedure. In order to prevent branch vessel occlusion, these branch vessels are typically stented with covered balloon expandable stents using standardized techniques.

SUMMARY:
The primary objective of the clinical investigation "Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Juxtarenal Aortic Aneurysms" is to assess the use of the Physician-Modified Endovascular Grafts to repair juxtarenal aneurysms in high-risk subjects considered to be unsuitable candidates for open surgical repair, have limited or no other options for treatment, and having appropriate anatomy. The primary intent of the study is to assess safety and preliminary effectiveness of the device:

* acutely (i.e., treatment success and technical success);
* at 30 days (i.e., the rate of major adverse events (MAE)); and
* at 6 months, 12 months and annually to 5 years (i.e., the proportion of treatment group subjects that achieve and maintain treatment success).

DETAILED DESCRIPTION:
The primary objective of the clinical investigation Physician Modified Endovascular Grafts for the Treatment of Elective, Symptomatic or Ruptured Juxtarenal Aortic Aneurysms is to assess the use of the Physician-Modified Endovascular Grafts to repair juxtarenal aneurysms in high-risk subjects considered to be unsuitable candidates for open surgical repair, have limited or no other options for treatment, and having appropriate anatomy. The primary intent of the study is to assess safety and preliminary effectiveness of the device acutely (i.e., treatment success and technical success), at 30 days (i.e., the rate of major adverse events (MAE)) and at 6 months, 12 months and annually to 5 years (i.e., the proportion of treatment group subjects that achieve and maintain treatment success).

ELIGIBILITY:
Inclusion Criteria:

All patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Patient is ≥ 18 years of age
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study)
3. Patient or Legally Authorized Representative has signed an Institutional Review Board (IRB) approved Informed Consent Form
4. Patient has a juxtarenal abdominal aortic aneurysm that meets at least one of the following:

   1. An aneurysm with a maximum diameter of ≥ 5.5 cm for male (≥ 5.0 cm for female) or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
   2. Aneurysm with a history of growth > 0.5 cm in 6 months
   3. Saccular aneurysm deemed at significant risk for rupture
   4. Symptomatic aneurysm
   5. Ruptured aneurysm
5. Patient has patent iliac or femoral arteries, with or without the use of conduit, that will allow endovascular access with the physician modified endovascular graft.
6. Patient has a suitable non-aneurysmal proximal aortic neck of ≥ 2 mm inferior to the most distal renal artery ostium.
7. Patient has a suitable non-aneurysmal distal iliac artery length (seal zone) of ≥ 15mm. The resultant repair should preserve patency in at least one hypogastric artery.
8. Patient has a suitable non-aneurysmal proximal aortic neck diameter between 20 and 32 mm, averaged across the diameters at the Celiac, SMA, at the lowest patent renal artery and at the midpoint of the renal arteries.
9. Patient has suitable non-aneurysmal distal common iliac diameters between 8 and 20 mm.
10. Patient has juxtarenal aortic neck angulation ≤ 60°
11. Target branch vessel diameter ≥ 5 mm.
12. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

Patients that meet ANY of the following are not eligible for enrollment into the study:

1. Patient has a mycotic aneurysm or has an active systemic or local infection that may increase the risk of endovascular infection
2. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina)
3. Patient has a major surgical or interventional procedure, not related to the endovascular repair, planned within +/- 30 days of the AAA repair.
4. Patient has history of an aortopathic connective tissue disease (e.g. Marfan's or Ehler's-Danlos syndrome).
5. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
6. Patient has known allergy or intolerance to stainless steel, nitinol or gold (gold-coated tungsten).
7. Patient has a body habitus that would inhibit X-ray visualization of the aorta
8. Patient has a limited life expectancy of less than 1 year
9. Patient is currently participating in another investigational device or drug clinical trial
10. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pretreatment, required treatment, and post-treatment procedures and evaluations.
11. Thrombus or excessive calcification within the neck of the aneurysm
12. Branch vessel stenosis ≥ 80%
13. Patient treatable on label with FDA approved EVAR or FEVAR device and can wait for device availability.
14. Subject is willing and eligible to enroll in a manufacturer-sponsored study at the investigational site, or the subject is willing and eligible to participate in a study with a manufacturer-made device at another institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events | Up to 30 days
  The proportion of patients that experience a rate of Major Adverse Events
Effectiveness | Up to 12 months
  Technical Success, defined as successful delivery and deployment of the physician modified endovascular graft with preservation of those branch vessels intended to be preserved.
  * Freedom from Type I & III endoleaks
  * Freedom from stent graft migration
  * Freedom from abdominal aortic aneurysm enlargement
  * Freedom from Aortic aneurysm rupture and conversion to open repair

SECONDARY OUTCOMES:
Occurrence of the safety events | Up to 5 years
  * Mortality
  * Aneurysm related mortality
  * Aneurysm rupture
  * Major Adverse Events
  * Renal failure with or without permanent dialysis
  * Graft infection
Technical Success | Up to 30 days
  Technical Success is a composite of the following:
  * Successful access to the arterial system using remote arterial exposure, percutaneous technique, or open surgical conduits
  * Successful delivery and deployment at the intended implantation site
  * Successful side branch catheterization and placement of bridging stents with restoration and maintenance of flow in all intended target vessels
  * Successful withdrawal of the delivery system
  * Patency of all endovascular graft and stent components
  * Absence of device deformations requiring unplanned placement of an additional device
  * Absence of Type I and III endoleaks at completion angiography
Stent Graft Migratoin | Up to 5 years
  Occurrence of stent graft migration >10 mm
All Endoleaks | Up to 5 years
  Occurrence of endoleaks (all types, including Type I and III)
AAA Enlargement | Up to 5 years
  Occurrence of AAA enlargement
Patency Related Events | Up to 5 years
  Occurrence of patency related events
Device Integrity Failure | Up to 5 years
  Occurrence of device integrity failure
Conversion to Open Repair | Up to 5 years
  Occurrence of Conversion to open repair
Secondary Intervention | Up to 5 years
  Occurrence of Secondary intervention (reason and type)

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Lyden, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No